CLINICAL TRIAL: NCT07244809
Title: Probing the Role of Mitochondrial Oxidative Stress in Impaired Vascular Function Among Young Adults With Early Life Adversity
Acronym: PROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: MitoQ Limited (Unknown)
Responsible Party: Principal Investigator, Nathaniel Jenkins, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202504919
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Adverse Childhood Experience; Endothelial Function (FMD); Endothelial Injury; Mitochondrial Function; Oxidative Stress; Psychosocial Influence on Cardiovascular Disease
Keywords: flow mediated dilation; mitoquinone mesylate; placebo; early life adversity; trier social stress test
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitoquinone Mesylate (MitoQ) (Experimental): Mitoquinone Mesylate (160 mg, single dose)
  Interventions: Dietary Supplement: Mitoquinone mesylate (MitoQ)
- Placebo (Placebo Comparator): Matched placebo (microcrystalline cellulose and tapioca, 160 mg, single dose)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mitoquinone mesylate (MitoQ) — Participants will consume a single 160 mg dose of mitoquinone mesylate, provided in the form of 6, 20 mg capsules, with water.
  Arms: Mitoquinone Mesylate (MitoQ)
Dietary Supplement: Placebo — Participants will consume a single 160 mg dose of microcrystalline cellulose and tapioca (placebo), provided in 20 mg capsules, with water.
  Arms: Placebo

SUMMARY:
Adverse childhood experiences (ACEs) represent highly stressful events in the first 18 years of life that include abuse, neglect, and household and community-level dysfunction. Greater exposure to ACEs are associated with greater increases in the risk of cardiovascular diseases and death. Our laboratory has previously observed that vascular function is disrupted in young adults with prior ACE exposure, even though these individuals appear to be healthy clinically (i.e., no classic clinical cardiovascular disease risk factors). There is a need to identify and understand the biological mechanisms underlying these vascular impairments to inform effective interventions to reduce cardiovascular risks the millions of individuals affected by ACEs.

The body's response to stress is coordinated across various systems, all of which depend on energy supplied by mitochondria (often referred to as the "powerhouse of cells"). Based on new evidence across multiple physiological systems from our team, our overarching hypothesis is that disruption of mitochondrial function contributes to cardiovascular impairments among young adults with ACEs. Here we propose the initial pilot work necessary to begin to understand these associations, which will directly inform identification of individuals who may be most vulnerable to stress-related cardiovascular risk and the development of interventions to promote cardiovascular-stress resilience.

Our aims are to:

1. Determine whether mitochondrial oxidative stress contributes to impaired vascular function among young adults who experienced early life adversity.
2. Determine whether reducing mitochondrial oxidative stress improves the cellular stress and integrated cardiovascular response to laboratory-based psychosocial stress among young adults who experienced early life adversity.

DETAILED DESCRIPTION:
Adverse childhood experiences (ACEs) represent highly stressful events in the first 18 years of life that include abuse, neglect, and household and community-level dysfunction. ACEs promote cardiovascular morbidity and mortality in a graded, dose-dependent manner1 and are thus a significant, widespread determinant of cardiovascular disease (CVD). In agreement with preclinical evidence,2 we have established that young adults (18-29 y) with prior ACE exposure exhibit impaired vascular endothelial function (VEF)3 as evidenced by reduced flow mediated dilation even in the absence of clinical CVD risk factors. The vascular endothelium is a regulatory organ that plays a critical role in maintaining cardiovascular homeostasis, and our findings indicate that vascular endothelial dysfunction is one of the earliest identifiable pathophysiological mechanisms linking ACE exposure with future CVD. There remains a critical biomedical need to identify and understand the psychobiological mechanisms underlying ACEs-related vascular endothelial dysfunction to inform effective interventions to improve cardiovascular health in the millions of individuals affected by ACEs. The physiologic response to stress is coordinated across various physiological systems, all of which depend on energy supplied at the cellular level by mitochondria. Based on novel evidence across multiple physiological systems from our team, our overarching hypothesis is that dysregulation of mitochondrial function due to chronic stress burden - or mitochondrial allostatic load (MAL) - promotes dysregulation of the physiological stress response which is ultimately transduced to impairments in VEF in young adults with ACEs. Notably, our preliminary evidence also suggests that psychological resilience and executive functions such as cognitive reappraisal may moderate these relations, reducing MAL and preserving VEF in the face of substantial adversity. Here we propose the critical work necessary to understand these associations, which will directly inform identification of individuals who may be most vulnerable to stress-related cardiovascular risk and the development of interventions to promote cardiovascular-stress resilience.

In this study, we will use an acute dose of a mitochondrial targeted antioxidant supplement (MitoQ; or placebo) to experimentally interrogate the role of mitochondrial oxidative stress is associated with improvements in 1) vascular endothelial function and 2) cellular and integrated cardiovascular responses to a standardized laboratory based psychosocial stressor in young adults with Adverse Childhood Experiences.

Participants will report to the laboratory, provide a blood sample and have vascular endothelial function assessed using a specialized test known as flow mediated dilation, consume a single acute dose of MitoQ previously demonstrated to be effective and safe for acutely decreasing mitochondrial oxidative stress in humans OR placebo, and then have vascular endothelial function measured again. Next, participants will provide another blood sample before undergoing a standardized and commonly used laboratory psychosocial stress test known, before providing additional blood samples after test completion.

1. Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, et al. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults: The adverse childhood experiences (ace) study. American Journal of Preventive Medicine. 1998;14:245-58. 2. Su S, Jimenez MP, Roberts CT, Loucks EB. The role of adverse childhood experiences in cardiovascular disease risk: A review with emphasis on plausible mechanisms. Curr Cardiol Rep. 2015;17:88. PMC4941633 3. Jenkins NDM, Rogers EM, Banks NF, Tomko PM, Sciarrillo CM, Emerson SR, Taylor A, et al. Childhood psychosocial stress is linked with impaired vascular endothelial function, lower sirt1, and oxidative stress in young adulthood. Am J Physiol Heart Circ Physiol. 2021;321:H532-H41. PMC8461842

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years
* ACE score >=4

Exclusion Criteria:

* Resting arterial blood pressure >140/90 mmHg
* BMI <=17 or >= 35
* Are on a weight-loss diet or involved in a formal weight-loss program or are not intentionally weight stable for 6 months (+/- 5 kg) prior to the study.
* Cardiovascular or metabolic prescription drug use
* Vasoactive antidepressant drug use (SSRIs and clonidine)
* Current heavy alcohol use, as defined as binge drinking on 5 or more days in the last month, or consuming more than 7 (women) or 14 (men) drinks per week in the last month (per NIAAA definition)
* Current or recent (within the last 6 mo.) illicit drug use disorder as indicated by a score of 3 or greater on the Drug Abuse Screening Test (DAST-10)
* Current tobacco or nicotine use
* Vaping
* Regular vigorous (>6 METs) aerobic exercise (>4 bouts/week, >30 min/bout)
* dietary supplementation with antioxidants or habitual use of NSAIDs
* Currently pregnant or breastfeeding

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular endothelial function | Prior to supplementation and 60 minutes after supplementation
  Vascular endothelial function will be assessed using the brachial artery flow mediated dilation technique
Blood pressure | 75 minutes after supplementation, during, and for 45 minutes after completion of the Trier Social Stress Test.
  The blood pressure response to psychosocial stress induced by the Trier Social Stress Test will be determined using beat-to-beat blood pressure measurement by finger photoplethysmography (or brachial artery blood pressure in the case of equipment errors). The Trier Social Stress Test will be performed after post-supplementation measurement of vascular endothelial function (FMD).
Endothelial Cell Microparticle Release | 60 minutes after supplementation and immediately following, 5-10 min, 15-20 min, and 45 min following the Trier Social Stress Test.
  Endothelial cell microparticle release will be quantified from platelet-poor plasma in response to psychosocial stress induced by the Trier Social Stress Test. The Trier Social Stress Test will be performed after post-supplementation measurement of vascular endothelial function (FMD).
Cortisol | 60 minutes after supplementation and immediately following, 5-10 min, 15-20 min, and 45 min following the Trier Social Stress Test.
  Cortisol will be quantified from drool collected passively to assess the HPA-axis response to psychosocial stress induced by the Trier Social Stress Test. The Trier Social Stress Test will be performed after post-supplementation measurement of vascular endothelial function (FMD).

SECONDARY OUTCOMES:
Total Peripheral Resistance | 75 minutes after supplementation, during, and for 45 minutes after completion of the Trier Social Stress Test.
  The total peripheral resistance response to psychosocial stress induced by the Trier Social Stress Test will be determined using beat-to-beat blood pressure measurement by finger photoplethysmography. The Trier Social Stress Test will be performed after post-supplementation measurement of vascular endothelial function (FMD).
Cardiac Output | 75 minutes after supplementation, during, and for 45 minutes after completion of the Trier Social Stress Test.
  The cardiac output response to psychosocial stress induced by the Trier Social Stress Test will be determined using beat-to-beat blood pressure measurement by finger photoplethysmography using ModelFlow. The Trier Social Stress Test will be performed after post-supplementation measurement of vascular endothelial function (FMD).
Growth Differentiation Factor 15 | 60 minutes after supplementation and immediately following, 5-10 min, 15-20 min, and 45 minutes after completion of the Trier Social Stress Test.
  Induction of GDF-15 will be quantified from plasma in response to psychosocial stress induced by the Trier Social Stress Test. The Trier Social Stress Test will be performed after post-supplementation measurement of vascular endothelial function (FMD).

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Laboratory of Applied Physiology and Lifestyle Medicine, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pilgrim JA, Crawford M. Low blood pressure and wellbeing. BMJ. 1993 Mar 6;306(6878):655. doi: 10.1136/bmj.306.6878.655-a. No abstract available. PMID 8461842
- [Background] Manson W, Annan WD. The structure of a phosphopeptide derived from -casein. Arch Biochem Biophys. 1971 Jul;145(1):16-26. doi: 10.1016/0003-9861(71)90004-x. No abstract available. PMID 4941633
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069